CLINICAL TRIAL: NCT00116883
Title: A Randomized, Double-blind, Parallel Group, Placebo Controlled, 6-week Study of the Effect of GW685698X Aqueous Nasal Spray 100mcg QD on the Hypothalamic Pituitary Adrenocortical (HPA) Axis in Children 2 to 11 Years of Age With Perennial Allergic Rhinitis (PAR).
Brief Title: A Study Of GW685698X For The Treatment Of Perennial Allergic Rhinitis In Pediatrics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR100012
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: GW685698X; perennial allergic rhinitis; pediatric; intranasal corticosteroid; HPA axis function
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: GW685698X aqueous nasal spray

INTERVENTIONS:
Drug: GW685698X aqueous nasal spray

SUMMARY:
The purpose of this study is to assess the effect of an aqueous nasal spray investigational compound GW685698X compared to placebo on the hypothalamic pituitary adrenocortical (HPA) axis system in children 2 to 11 years of age with perennial allergic rhinitis.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis and history of perennial allergic rhinitis.
* Must be willing to stay overnight in the clinic at the beginning and end of the study for the collection of urine and blood samples over 24 hours.
* Must comply with all study procedures and be literate.

Exclusion criteria:

* Significant concurrent medical conditions.
* Certain medications such as corticosteroids and allergy medications.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2005-02; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
HPA axis function at baseline and after 6 weeks of treatment as measured by 24 hour urine and serial serum cortisol assessments in domiciled subjects

SECONDARY OUTCOMES:
Results of adverse event, laboratory, nasal examination, vital sign, ECG and pharmacokinetic assessments.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (12):
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: FFR100012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR100012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR100012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR100012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR100012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR100012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR100012 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register